CLINICAL TRIAL: NCT02719431
Title: Drug-Drug Interaction Study to Assess the Effects of Multiple-Dose Administration of K-877 on the Pharmacodynamics and the Pharmacokinetics of Multiple-Dose Administration of Warfarin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: K-877-108
Record Dates: First submitted 2016-01-29; First posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
MeSH Terms: interventions — Warfarin; K-877 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Warfarin/Warfarin + K-877 (Other)
  Interventions: Drug: Warfarin; Drug: K-877

INTERVENTIONS:
Drug: Warfarin
Drug: K-877

SUMMARY:
The purpose of this study is to assess the effects of K-877 on the pharmacodynamics and the pharmacokinetics of warfarin in healthy adults volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides written informed consent before any study specific evaluation is performed.
* Subject is a healthy adult male or female volunteer between the ages of 18 and 45 years, inclusive.
* Subject has a body mass index of 18 to 30 kg/m², inclusive.

Exclusion Criteria:

* Subject has clinically relevant abnormalities in the screening or check in assessments.
* Subject has clinically significant out-of-range PT, INR, activated partial thromboplastin time, fibrinogen, protein C, or protein S.
* Subject has abnormal prolongation of skin bleeding time at Screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
International normalized ratio (INR) | 22 Days

CONTACTS AND LOCATIONS:
Locations (1):
- Austin, Texas, United States